CLINICAL TRIAL: NCT06431139
Title: Intensive Physical Exercise Versus Standard Exercise During Rehabilitation of Patients With Traumatic Brain Injury - a Randomised Pilot and Feasibility Trial
Brief Title: Intensive Physical Exercise Versus Standard Exercise During Rehabilitation of Patients With Traumatic Brain Injury
Acronym: INSPIRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Riberholt (Other)
Responsible Party: Sponsor-Investigator, Christian Riberholt, Head of therapy and senior researcher, PT, MR, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-24001505
Record Dates: First submitted 2024-05-07; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Intensive exercise; Rehabilitation; Randomised trial; Feasibility; Pilot; Sit-to-stand exercise
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The trial will use assessors blinded to the allocation and in charge of testing the following outcomes: 30 seconds chair stand test, 10-meter walk test, 6-minute walking test, and the Montreal Cognitive Assessment Scoring (MoCA) Two statisticians that will perform the statistical analysis are blinded to the allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INSPIRE group (Experimental): Intervention group. Daily intensive sit-to-stand exercises following a described algorithm and utilising motor-relearning principles of feedback to increase the participant's motivation. This exercise is an addition to standard care.
  Interventions: Other: INSPIRE intervention protocol
- Standard care group (No Intervention): Treatment in this group will be standard care interventions performed at the rehabilitation department.

INTERVENTIONS:
Other: INSPIRE intervention protocol — 2-week training program with daily sit-to-stand exercises. Each working day the participant's goals will be adjusted, until exercising a minimum of 100 repetitions using an exercise progression table. When participants complete one level, they will progress to the next level the following day. Participants who do not reach the goals at level one will continue to strive to reach the 100 repetitions. The number of repetitions can be split and performed throughout the day. As the participants' capacity for doing the exercises increases, so will the number of repetitions within each bout of sit-to-stand. Participants are allowed to do the number of repetitions from a higher exercise level if they can and will continue by progressing from that level on the next day. The repetitions will be done from a height that makes it possible to accomplish the sit-to-stand movement. Therefore, the height of the sitting surface will be adjusted according to the participant's abilities.
  Arms: INSPIRE group

SUMMARY:
The aim of this randomised multicentre clinical feasibility and pilot trial is to test if a sit-to-stand trial protocol is feasible regarding the increased intensity, trial recruitment, and completion of outcome data in patients with moderate to severe traumatic brain injury during the rehabilitation phase. For the trial to be feasible, all outcomes must be achieved.

The primary hypothesis is that it is feasible to progressively increase the number of repetitions of sit-to-stand exercises in patients with moderate to severe traumatic brain injury admitted to a rehabilitation department during the intervention period.

Furthermore, the investigators hypothesize that the increased number of repetitions will increase the participant's functional capabilities regarding sit-to-stand and walking, decrease resting heart rate, blood pressure, and metabolism, reduce inflammatory and brain injury biomarkers, and improve the cognitive performance.

DETAILED DESCRIPTION:
This is a randomised multicentre clinical feasibility and pilot trial, where assessors and statisticians will be blinded. Forty-four participants with moderate to severe traumatic brain injury will be randomised to INSPIRE versus standard care as soon as they are able to understand and execute simple commands twice during one day. Participants in the INSPIRE group will undergo two weeks of intensive sit-to-stand exercise using an algorithm to increase the intensity daily. The trial uses predefined dose-limiting events to reduce training intensity in participants experiencing exercise-related adverse events that limit other daily activities and rehabilitation (e.g. muscle soreness and pain). Overall feasibility will be assessed by determining the inclusion rate, exercise completion rate, and completion of the Glasgow Outcome Scale - Extended. As exploratory clinical outcomes, the investigators will assess serious adverse events and adverse events not considered serious, physical function, cardiovascular and metabolic health, fatigue, and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe traumatic brain injury with Glasgow Coma Score <13 within the first 24 hours (ICD10, DS06)
* Admitted for rehabilitation at the Department of Brain and Spinal Cord Injury, Division of Brain Injury, Rigshospitalet, the Regional Hospital, Hammel Neurocentre or the Acquired Brain Injury Rehabilitation Centre, Alfred Hospital
* 18 years old or older
* Patients (or next of kin) should be able to understand written and spoken Danish or English to consent to participation in the trial validly
* Specifically for Australian participants: eligibility for Medicare

Exclusion Criteria:

* Unstable fractures of the lower extremities
* Amputation of lower extremity
* Spinal cord injury
* Total paralysis of both lower extremities
* Agitated or combative behaviour
* Diagnosed with a progressive neurological disorder (e.g. Alzheimer's, Parkinson's disease, multiple sclerosis) prior to traumatic brain injury, as it could potentially interfere with serum biomarker levels
* Previous structural brain injury (e.g. stroke or brain surgery)
* No valid consent from the participant or next of kin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of sit-to-stand | during the intervention
  The difference in the number of sit-to-stand performed in the INSPIRE group compared to the control group using linear regression during the two-week intervention period.

SECONDARY OUTCOMES:
The number of participants included in the trial | 1,5 years
  Of all eligible patients, at least 76% (95% CI 63% to 86%, 1-sample proportions test with continuity correction) must consent (by themselves or by proxy) to inclusion in the trial, corresponding to 44/58 eligible patients included
Participants completing GOSE | 6 months, 1 year
  The number of participants completing the Glasgow Outcome Scale extended at six months and one year must be above 89% (95% CI 76% to 96%), corresponding to 40/44 participants.

OTHER OUTCOMES:
Dose-limiting events | during the intervention, 72-hours after end of intervention
  Examples of this could be fatigue or muscle pain that limits the participant in other activities of daily living and thereby reduces their amount of other rehabilitation services during the day
Glasgow Outcome Scale - Extended | at discharge, 6 months, 1 year
  The scale is a global scale evaluating the independent function after traumatic brain injury.
Number of sit-to-stand exercises in each group during the intervention period (continuous outcome) | during the intervention
  The total number of sit-to-stands in each group will be measured using an activity monitor placed on the participant's sternum and hip (Sens motion®, Copenhagen, Denmark)
Number of sit-to-stand exercises during the 30-second chair stand test (continuous outcome) | Baseline, 1 day after the intervention
  The test is administered using a stopwatch and a chair. The participant is instructed to do sit-to-stand movements for 30 seconds. Time begins when the participant initiates the movement.
Walkers and non-walker (dichotomous outcome) | Baseline, 1 day after the intervention
  Walkers are defined by the ability to walk at any pace, with any walking aid, over minimum 50 meters independently (i.e. independent from physical assistance).
10-meter walk test (continuous outcome) | Baseline, 1 day after the intervention
  The walkers in each group will undergo a 10-meter walk test to assess walking speed
6-minute walking test (continuous outcome) | Baseline, 1 day after the intervention
  The walkers in each group will undergo a 6-minute walking test to assess and endurance
Resting blood pressure | Baseline, 1 day after the intervention
  Resting blood pressure will be measured on both arms for 5 minutes continuously before the first training session (8 am) using photoplethysmography to measure beat-to-beat blood pressure non-invasively.
Resting heart rate | Baseline, 1 day after the intervention
  An ordinary electrocardiogram available at the respective departments will be used to measure resting heart rate.
Blood samples | Baseline, 1 day after the intervention
  The blood samples will be analysed for high-sensitivity C-reactive protein, neutrophil-to-lymphocyte ratio, HbA1c, blood glucose, c-peptide insulin, blood lipids, inflammatory biomarkers, neuronal cell injury biomarkers, astroglia cell injury biomarkers, and axonal injury biomarkers. Finally, biomarkers associated with subacute/chronic traumatic brain injury phase will be analysed.
The Montreal Cognitive Assessment (MoCA) | Baseline, 1 day after the intervention, 6 months, 1 year
  The MoCA is a short cognitive questionnaire designed to test for mild cognitive impairments.
Fatigue severity scale (FSS) | Baseline, 1 day after the intervention, 6 months, 1 year
  The Fatigue Severity Scale examines the severity of fatigue with a 9-item scale, and how it can affect a person's daily lifestyle when they have a chronic disease/disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Christian G Riberholt, PT, MR, PhD, Study Director — Dept. of Brain and Spinal Cord Injury, Division of Brain Injury, Copenhagen University Hospital - Rigshospitalet; Christina G Kruuse, Professor, Study Director — Dept. of Brain and Spinal Cord Injury, Division of Brain Injury, Copenhagen University Hospital - Rigshospitalet